CLINICAL TRIAL: NCT03321201
Title: Cauterization Versus ﬁbrin Glue for Conjunctival Autografting in Primary Pterygium Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Livia Puljak, Associate Professor, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTERYGIUM1
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pterygium of Conjunctiva and Cornea
MeSH Terms: conditions — Pterygium Of Conjunctiva And Cornea | interventions — Cautery; Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Surgeons will not be blinded. All the other investigators, as well as study participants, outcome assessors and author that will analyze the data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cauterization (Experimental)
  Interventions: Procedure: Cauterization
- Fibrin glue (Active Comparator)
  Interventions: Procedure: Fibrin glue

INTERVENTIONS:
Procedure: Cauterization — To ensure the stability of the graft during cuttings, four sealing wraps will be installed, which will be removed after cauterisation is completed. Autograft and conjunctiva will be approximated by surgical forceps and will be cauterized using a bipolar cutter (Erbe ICC 50) with a force 1-3 / 20. Forceps will be released slowly to prevent elevation of the graft. The same procedure will be performed 10 times until graft is well firmed. Graft stability will be checked up with a sponge and additional cauterization will be preformed if needed.
  Arms: Cauterization
Procedure: Fibrin glue — Fiber adhesive (Tissel 1 mL kit4-iu) will be prepared according to manufacturer's instructions. Preparation time will be approximately 10-15 min per kit. Once mixed the fibrin glue is usable up to 4 h. For the purpose of the study preparation of the fibrin glue will be performed by a nurse.
  Arms: Fibrin glue

SUMMARY:
Pterygium is a noncancerous growth of the conjunctival tissue over the cornea. It is a progressive disease that may lead to visual impairment in advanced stages, as well as restriction of ocular motility, chronic inflammation and cosmetic concerns. Surgical removal is the treatment of choice, but recurrence of pterygium is a frequent problem. In this randomized controlled cauterization will be compared with ﬁbrin glue for conjunctival autografting in primary pterygium surgery.

ELIGIBILITY:
Inclusion criteria:

* adults (older than 18 years of age)
* both sexes
* primary nasal pterygia ˃4 mm, which tends to increase, including patients with reduced visual acuity, chronic inflammation, cosmetic reasons
* if the patients had a bilateral pterygium, only one eye will be operated

Exclusion criteria:

* connective tissue disease
* prior eye surgery
* chronic use of topical drugs (anti-glaucoma drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pterygium | 180 days
  Any re-growth of tissue from the area of excision across the limbus onto the cornea.

SECONDARY OUTCOMES:
Surgical time | During the surgery
  Surgical time: total operational time required for completion of the operation (measured in minutes)
Complication rate | 7, 30 and 180 days
  Complication rate will be analyzed as the occurrence of at least one of the following major complications such as dehiscence, displacement or loss of the autograft, infection, haemorrhage, oedema, ﬁbrosis, retraction and other indications that required special treatment
Pterygium-induced astigmatism | 7, 30 and 180 days
  Measured as described by Hsu 2014
Ocular surface condition | 7, 30 and 180 days
  The Ocular Surface Disease Index (OSDI) is a 12-question validated questionnaire used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision. The OSDI scoring scale ranges from 0 to 100. The lower the score, the more symptomatic relief from dry eye symptoms a patient experiences. Baseline-adjusted scores were tabulated; a negative number change from baseline indicates a perceived improvement in ocular comfort.
Postoperative discomfort, tearing, pain and foreign body sensation | 7, 30 and 180 days
  Using modified scale from Lim Bon Siong et al: (0) none, no pain, (1) very mild, (2) mild, pain causing some discomfort, (3) moderate, pain that partially interferes with usual activity or sleep, (4) sever, pain that completely interferes with usual activity or sleep.
Pain | 7, 30 and 180 days
  Numerical rating scale (NRS) ranging from 0 to 10, where 0 = No pain and 10 = Pain as intense as you can imagine.
Economic Analysis | 180 days
  Cost of each intervention
Flap time | During the surgery
  Time needed for preparing and repositioning of the conjunctival grafts (measured in minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be made available to other researchers on request.

REFERENCES:
- [Derived] Lesin M, Paradzik M, Marin Lovric J, Olujic I, Ljubic Z, Vucinovic A, Bucan K, Puljak L. Cauterisation versus fibrin glue for conjunctival autografting in primary pterygium surgery (CAGE CUP): study protocol of a randomised controlled trial. BMJ Open. 2018 Jun 27;8(6):e020714. doi: 10.1136/bmjopen-2017-020714. PMID 29950464